CLINICAL TRIAL: NCT03935035
Title: Online PTSD Treatment for Young People and Carers - Case Series
Acronym: OPTYC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Medical Research Council (Other Government); South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MR/P017355/1
Record Dates: First submitted 2019-04-08; First posted 2019-05-02 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-04

CONDITIONS: Post Traumatic Stress Disorder
Keywords: adolescents; internet-delivered; online; young people; trauma; cognitive therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Uncontrolled case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- internet-Cognitive Therapy for PTSD (Experimental): This is a single-arm study. All participants will receive the same therapist supported, internet-delivered intervention.
  Interventions: Behavioral: internet-delivered Cognitive Therapy for PTSD (iCT)

INTERVENTIONS:
Behavioral: internet-delivered Cognitive Therapy for PTSD (iCT) — Participants will receive 10 hours of Cognitive Therapy for PTSD over 12 weeks, with a baseline assessment at the beginning and follow up interview at the end of treatment. The treatment consists of online modules (9 core modules, 11 optional modules and parent/carer modules) and a weekly phone call with a qualified and trained therapist.

SUMMARY:
Post Traumatic Stress Disorder (PTSD) is prevalent and impairing in children and young people. Effective face to face treatments exist, including Cognitive Therapy for PTSD (CT-PTSD), developed by the researchers' group. However, few young people access effective treatments.

The researchers are therefore developing a website and smart-phone App that will improve accessibility of this treatment by allowing trained therapists to deliver CT-PTSD over the internet (iCT) to young people (12-17 years old) with PTSD. This study aims to provide an initial evaluation of iCT. This will be done by running an uncontrolled case series with 6 young people.

The objectives of the case series are to: to gauge acceptability of the programme to young people, carers, and therapists; to measure adherence to the programme; to test the battery of measures for acceptability; and to obtain estimates of clinical change.

DETAILED DESCRIPTION:
PTSD is prevalent among young people, and is distressing and impairing. Face-to-face trauma-focussed CBT (TFCBT) is an effective short-term therapy for PTSD in young people. The researchers previously developed Cognitive Therapy for PTSD (CT-PTSD) in children and young people, and have shown in 2 published RCTs that it is efficacious when delivered face-to-face. However, most young people with PTSD do not receive effective, evidence-based treatments. This is in part due to under-capacity in NHS CAMHS, and in part due to the burden and inconvenience to young people in attending face-to-face appointments in a clinic. In this project the researchers propose to make CT for PTSD widely available to young people by delivering the therapy via the internet, with therapist support. The rationale for this approach is that (1) young people will engage with internet-delivered therapy, and online therapies for other disorders such as depression have demonstrated efficacy in clinical trials; (2) effective online therapies for adults with PTSD have been developed and evaluated; (3) no online treatments for young people with PTSD have yet been developed.

An uncontrolled case series will be run with N=6 young patients. Young people who are referred to the South London and Maudsley NHS Foundation Trust CAMHS service, and who meet the eligibility criteria, will be invited to take part in the case series. After both the young person and their carer or parent have provided informed consent (or assent), they will complete several baseline assessment measures. These measures will be completed at a face-to-face meeting in the Tier 4 National and Specialist Trauma, Anxiety and Depression (TAD) NHS clinic, and online. The young person and family will meet the young person's therapist face-to-face at this initial assessment meeting. After assessment, the young person that will be treated remotely using iCT for up to 12 weeks.

This treatment will include regular (at least weekly) telephone contact with the therapist, and other contact with the therapist during the week using a messaging function within the iCT App. The young person will be asked to complete a mood rating and a brief 8-item questionnaire about PTSD symptoms once a week during treatment: this mirrors what happens during standard face-to-face care in the TAD NHS clinic. At mid treatment, the young person will be asked to complete one additional 25-item questionnaire about thoughts related to trauma. Risk monitoring including monitoring of adverse events will be carried out during weekly phone calls.

Post treatment, the young person will attend the TAD NHS clinic for a face-to-face clinical interview and will complete a questionnaire pack online. At this meeting, the young person will complete feedback ratings on the acceptability of the design of online treatment modules using 4 simple 0-10 scales (about the overall design appeal, ease-of-use, comprehension, and likelihood of recommending the program to a friend with similar problems). The young person will be interviewed about their experience of using the iCT program (an "exit interview"). Acceptability of the questionnaire battery will be assessed by asking young people to complete an end-of-treatment rating using a 0-100 scale. The young people's parents or carers will also take part in a clinical interview about the young person, will complete a questionnaire pack online, and will be invited to take part in an interview about their experience as a parent or carer of using the iCT program.

N=6 young people will be treated as part of this case series. Young people's and their parents' qualitative feedback on the acceptability of the iCT programme will be reported using data from the exit interviews and from the acceptability rating scales. Averse events during therapy will also be reported. Reliable Clinical Change on a standardised questionnaire of PTSD symptoms (the CPSS-5) will be reported as a preliminary signal of clinical effect. Reliable Clinical Improvement is shown by a reduction of 8 points on the CPSS-5. Acceptability of the outcome measures will be gauged by scrutinising completion rates.

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged 12-17 years old
* Main presenting problem is PTSD and there is a not a co-morbid problem that would preclude treatment of PTSD.
* PTSD symptoms related to a single trauma
* Participant has access to compatible smartphone and larger computing device (e.g. laptop, desktop computer, iPad) with internet access.
* Participant is proficient in speaking and writing in the English language, sufficient to participate in treatment without an interpreter.

Exclusion Criteria:

* Brain damage assessed by clinical interview with parents / carers
* Intellectual disability assessed by clinical interview with parents / carers
* Pervasive developmental disorder or neurodevelopmental disorder assessed by clinical interview with parents / carers
* Other psychiatric diagnosis that requires treatment before PTSD, determined by clinical interview and questionnaires
* Moderate to high risk to self assessed in clinical interview
* Ongoing trauma-related threat assessed in clinical interview
* Started treatment with psychotropic medication, or changed medication, within the last 2 months, assessed in clinical interview
* Currently receiving another psychological treatment, assessed in interview
* Have already received Trauma Focused CBT in relation to the same traumatic event that the young person is currently seeking treatment for.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
PTSD symptom scale: Clinician Administered PTSD Scale for Children and Adolescents (CAPS-CA-5, Pynoos et al., 2015) | Baseline
  Clinician Administered. The time period covered is the past month. Items are rated 0-4 based on frequency and severity of symptoms (0=absent, 1= mild, 2=moderate, 3 = severe, 4 = extreme). PTSD diagnostic status is determined by first dichotomizing each symptom as "present" (if the symptom severity is rated 2 or higher) or "absent" (rated 0 or 1). Items pertain to the 4 criterion of PTSD outlined in the DSM-V; criterion B (items 1-5), criterion C (items 6-7), criterion D (items 8-14) and criterion E (items 15-20). PTSD may be diagnosed if the young person has at least one criterion B, one criterion C, two criterion D and two criterion E symptoms and if the disturbance has lasted for more than one month and causes clinically significant distress or functional impairment.
PTSD symptom scale: using the Clinician Administered PTSD Scale for Children and Adolescents (CAPS-CA-5, Pynoos et al., 2015) | post-intervention (at 4 months)
  Clinician Administered. The time period covered is the past month. Items are rated 0-4 based on frequency and severity of symptoms (0=absent, 1= mild, 2=moderate, 3 = severe, 4 = extreme). PTSD diagnostic status is determined by first dichotomizing each symptom as "present" (if the symptom severity is rated 2 or higher) or "absent" (rated 0 or 1). Items pertain to the 4 criterion of PTSD outlined in the DSM-V; criterion B (items 1-5), criterion C (items 6-7), criterion D (items 8-14) and criterion E (items 15-20). PTSD may be diagnosed if the young person has at least one criterion B, one criterion C, two criterion D and two criterion E symptoms and if the disturbance has lasted for more than one month and causes clinically significant distress or functional impairment.
PTSD symptoms: Child Post Traumatic Stress Scale (CPSS-5; Foa et al. 2001) | Baseline
  A self-report questionnaire with 27 items relating to the past one month. The first 20 items evaluate the frequency and severity of PTSD symptoms. Items are rated on a 5-point scale (0= not at all, 1 = <once a week, 2= 2-3 times per week, 3 = 4-5 times a week, 4 = 6 or more times per week). The final 7 items evaluate functional impairment an are scored 1 ('Yes') or 0 ('No') with scores ranging from 0-7, greater scores indicate greater impairment. From the first part of the CPSS scores can range between 0-80 with higher scores indicating greater symptom severity. A score of 31 or higher indicates PTSD.
PTSD symptoms: Child Post Traumatic Cognitions Inventory (CPTCI, McKinnon et al 2016) | Baseline
  A self-report questionnaire with 10 items. The CPTCI measures PTSD symptoms since the traumatic event occurred, on a scale of 1-4 (1= don't agree at all, 2 = don't agree a bit, 3 = agree a bit, 4 = agree a lot). Scores range from 0-40 with greater scores indicating greater symptom severity. A total score of 16 or above is considered clinically significant.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al 2005) | Baseline
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Child Post Traumatic Cognitions Inventory (CPTCI, McKinnon et al 2016) | Mid-Treatment (at 6 weeks)
  A self-report questionnaire with 10 items. The CPTCI measures PTSD symptoms since the traumatic event occurred, on a scale of 1-4 (1= don't agree at all, 2 = don't agree a bit, 3 = agree a bit, 4 = agree a lot). Scores range from 0-40 with greater scores indicating greater symptom severity. A total score of 16 or above is considered clinically significant.
PTSD symptoms: Child Post Traumatic Stress Scale (CPSS-5; Foa et al. 2001) | Post-treatment (at 4 months)
  A self-report questionnaire with 27 items relating to the past one month. The first 20 items evaluate the frequency and severity of PTSD symptoms. Items are rated on a 5-point scale (0= not at all, 1 = <once a week, 2= 2-3 times per week, 3 = 4-5 times a week, 4 = 6 or more times per week). The final 7 items evaluate functional impairment an are scored 1 ('Yes') or 0 ('No') with scores ranging from 0-7, greater scores indicate greater impairment. From the first part of the CPSS scores can range between 0-80 with higher scores indicating greater symptom severity. A score of 31 or higher indicates PTSD.
PTSD symptoms: Child Post Traumatic Cognitions Inventory (CPTCI, McKinnon et al 2016) | Post-treatment (at 4 months)
  A self-report questionnaire with 10 items. The CPTCI measures PTSD symptoms since the traumatic event occurred, on a scale of 1-4 (1= don't agree at all, 2 = don't agree a bit, 3 = agree a bit, 4 = agree a lot). Scores range from 0-40 with greater scores indicating greater symptom severity. A total score of 16 or above is considered clinically significant.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al 2005) | Post-treatment (at 4 months)
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al 2005) | 10-month follow up
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Child Post Traumatic Stress Scale (CPSS-5; Foa et al. 2001) | 10-month follow up
  A self-report questionnaire with 27 items relating to the past one month. The first 20 items evaluate the frequency and severity of PTSD symptoms. Items are rated on a 5-point scale (0= not at all, 1 = <once a week, 2= 2-3 times per week, 3 = 4-5 times a week, 4 = 6 or more times per week). The final 7 items evaluate functional impairment an are scored 1 ('Yes') or 0 ('No') with scores ranging from 0-7, greater scores indicate greater impairment. From the first part of the CPSS scores can range between 0-80 with higher scores indicating greater symptom severity. A score of 31 or higher indicates PTSD.
PTSD symptoms: Child Post Traumatic Cognitions Inventory (CPTCI, McKinnon et al 2016) | 10-month follow up
  A self-report questionnaire with 10 items. The CPTCI measures PTSD symptoms since the traumatic event occurred, on a scale of 1-4 (1= don't agree at all, 2 = don't agree a bit, 3 = agree a bit, 4 = agree a lot). Scores range from 0-40 with greater scores indicating greater symptom severity. A total score of 16 or above is considered clinically significant.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 1
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 2
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 3
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 4
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 5
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 6
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 7
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 8
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 9
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 10
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 11
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
PTSD symptoms: Children's Revised Impact of Event Scale (CRIES; Perrin et al., 2005) | Week 12
  A self-report questionnaire with 8 items (4 measuring intrusions, 4 measuring avoidance). The items assess symptoms over the past 7 days on a 4-point scale (0=not at all, 1= rarely, 3=sometimes, 5=often). Intrusion sub-scale is the sum of items 1,3,6 and 7. Avoidance sub-scale is the sum of items 2,4,5 and 8. Scores can range from 0-40 with greater scores indicating greater symptom severity. A total score of 17 or higher indicates PTSD.
Acceptability of iCT: Qualitative interviews | Post-Treatment (at 4 months)
  Qualitative interviews with N=6 young people, their carers, and their therapists.
Acceptability of iCT: Likert Scales | Post-Treatment (at 4 months)
  Young people will be asked to complete ratings of acceptability on a scale from 0 to 100.
Adherence to online intervention: time spent logged in to programme | up to week 12
  Time spent logged on to online programme in seconds:minutes:hours according to the device used (smartphone, tablet or computer).
Adherence to online intervention: number of times logged on | up to week 12
  The number of times a participant logs on to the online programme
Adherence to online intervention: number of modules completed | up to week 12
  The number of online modules the young person completes during the 12 week intervention
Adherence to online intervention: number of phone calls between therapist and young person | up to week 12
  The number of times the participant spoke to the therapist on the phone
Adherence to online intervention: time spent on phone calls with the therapist | up to week 12
  Time spent on phone calls with the therapist in seconds:minutes:hours
Adherence to online intervention: number of messages exchanged with the therapist | up to week 12
  Number of messages exchanged between the patient and the therapist

SECONDARY OUTCOMES:
Revised Children's Anxiety and Depression Scale (RCADS-C; Chorpita & Ebesutani 2014): Measure of young person's anxiety and depression symptoms | Baseline
  A 47-item self-report questionnaire. Items are rated on a 4-point scale (0= never, 1 = sometimes, 2= often, 3 = always). The RCADS can be scored using spreadsheets available from the developer. The young person's school year must be entered (enter the year number according to the US grade system) and a 't-score' is calculated. A t-score of 70 or more is considered clinically significant. The greater the t-score the greater the symptoms.
Revised Children's Anxiety and Depression Scale (RCADS-P Chorpita & Ebesutani 2014): Measure of young person's anxiety and depression symptoms | Baseline
  A 47-item parent rated questionnaire. Items are rated on a 4-point scale (0= never, 1 = sometimes, 2= often, 3 = always). The RCADS-P can be scored using spreadsheets available from the developer. The young person's school year must be entered (enter the year number according to the US grade system) and a 't-score' is calculated. A t-score of 70 or more is considered clinically significant. The greater the t-score the greater the symptoms.
Revised Children's Anxiety and Depression Scale (RCADS-C; Chorpita & Ebesutani 2014): Measure of young person's anxiety and depression symptoms | post-treatment (at 4 months)
  A 47-item self-report questionnaire. Items are rated on a 4-point scale (0= never, 1 = sometimes, 2= often, 3 = always). The RCADS can be scored using spreadsheets available from the developer. The young person's school year must be entered (enter the year number according to the US grade system) and a 't-score' is calculated. A t-score of 70 or more is considered clinically significant. The greater the t-score the greater the symptoms.
Revised Children's Anxiety and Depression Scale (RCADS-P Chorpita & Ebesutani 2014): Measure of young person's anxiety and depression symptoms | post-treatment (at 4 months)
  A 47-item parent rated questionnaire. Items are rated on a 4-point scale (0= never, 1 = sometimes, 2= often, 3 = always). The RCADS-P can be scored using spreadsheets available from the developer. The young person's school year must be entered (enter the year number according to the US grade system) and a 't-score' is calculated. A t-score of 70 or more is considered clinically significant. The greater the t-score the greater the symptoms.
Revised Children's Anxiety and Depression Scale (RCADS-C; Chorpita & Ebesutani 2014): Measure of young person's anxiety and depression symptoms | at 10-month follow up
  A 47-item self-report questionnaire. Items are rated on a 4-point scale (0= never, 1 = sometimes, 2= often, 3 = always). The RCADS can be scored using spreadsheets available from the developer. The young person's school year must be entered (enter the year number according to the US grade system) and a 't-score' is calculated. A t-score of 70 or more is considered clinically significant. The greater the t-score the greater the symptoms.
Revised Children's Anxiety and Depression Scale (RCADS-P Chorpita & Ebesutani 2014): Measure of young person's anxiety and depression symptoms | at 10-month follow up
  A 47-item parent rated questionnaire. Items are rated on a 4-point scale (0= never, 1 = sometimes, 2= often, 3 = always). The RCADS-P can be scored using spreadsheets available from the developer. The young person's school year must be entered (enter the year number according to the US grade system) and a 't-score' is calculated. A t-score of 70 or more is considered clinically significant. The greater the t-score the greater the symptoms.
Strength & Difficulties Questionnaire (SDQ-P; Goodman, 2001): Measure of young person's emotional and behavioural difficulties | Baseline
  Parent rated questionnaire with 25 items. Items are rated on a 3-point scale (0=not true, 1=somewhat true, 2= certainly true). There are 5 sub-scales each with scores ranging from 0-10. The total difficulties score is calculated by summing 4 of the sub-scales to give a score between 0-40. A total difficulties score of 17 or above is considered clinically significant. The greater the total score, the greater the difficulties experienced.
Strength & Difficulties Questionnaire (SDQ-P; Goodman, 2001): Measure of young person's emotional and behavioural difficulties | post-treatment (at 4 months)
  Parent rated questionnaire with 25 items. Items are rated on a 3-point scale (0=not true, 1=somewhat true, 2= certainly true). There are 5 sub-scales each with scores ranging from 0-10. The total difficulties score is calculated by summing 4 of the sub-scales to give a score between 0-40. A total difficulties score of 17 or above is considered clinically significant. The greater the total score, the greater the difficulties experienced.
Strength & Difficulties Questionnaire (SDQ-P; Goodman, 2001): Measure of young person's emotional and behavioural difficulties | at 10-month follow up
  Parent rated questionnaire with 25 items. Items are rated on a 3-point scale (0=not true, 1=somewhat true, 2= certainly true). There are 5 sub-scales each with scores ranging from 0-10. The total difficulties score is calculated by summing 4 of the sub-scales to give a score between 0-40. A total difficulties score of 17 or above is considered clinically significant. The greater the total score, the greater the difficulties experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Smith, PhD, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - King's College London/ South London and Maudsley NHS Foundation Trust, London
  - University of East Anglia/ Norfolk and Suffolk NHS Foundation Trust, Norwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foa EB, Johnson KM, Feeny NC, Treadwell KR. The child PTSD Symptom Scale: a preliminary examination of its psychometric properties. J Clin Child Psychol. 2001 Sep;30(3):376-84. doi: 10.1207/S15374424JCCP3003_9. PMID 11501254
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] McKinnon A, Smith P, Bryant R, Salmon K, Yule W, Dalgleish T, Dixon C, Nixon RD, Meiser-Stedman R. An Update on the Clinical Utility of the Children's Post-Traumatic Cognitions Inventory. J Trauma Stress. 2016 Jun;29(3):253-8. doi: 10.1002/jts.22096. Epub 2016 May 18. PMID 27191657
- [Background] Perrin, S., Meiser-Stedman, R., & Smith, P. (2005). The Children's Revised Impact of Event Scale (CRIES): validity as a screening instrument for PTSD. Behavioural and Cognitive Psychotherapy, 33(4), 487-498.
- [Background] Pynoos, R. S., Weathers, F. W., Steinberg, A. M., Marx, B. P., Layne, C. M., Kaloupek, D. G., Schnurr, P. P., Keane, T. M., Blake, D. D., Newman, E., Nader, K. O., & Kriegler, J. A. (2015). Clinician-Administered PTSD Scale for DSM-5 - Child/Adolescent Version.
- See also: Link to Perrin, Meiser-Stedman, & Smith, (2005). The Children's Revised Impact of Event Scale (CRIES): validity as a screening instrument for PTSD — https://ueaeprints.uea.ac.uk/50579/1/Perrin_et_al_2005_BCP_postprint.pdf
- See also: Link to Pynoos et al., (2015). Clinician-Administered PTSD Scale for DSM-5 - Child/Adolescent Version — https://www.ptsd.va.gov/professional/assessment/documents/CAPS-CA-5.pdf
- See also: Chorpita, B. F., Ebesutani, C., & Spence, S. H. (2014). Revised children's anxiety and depression scale user's guide. Unpublished Users Guide, University of California, Los Angeles. http://www. childfirst. ucla. edu/RCADSUsersGuide20140711.pdf. — https://scholar.google.co.uk/scholar?hl=en&as_sdt=0%2C5&q=Chorpita%2C+B.+F.%2C+Ebesutani%2C+C.%2C+%26+Spence%2C+S.+H.+%282014%29.+Revised+children%E2%80%99s+anxiety+and+depression+scale+user%E2%80%99s+guide.+Unpublished+Users+Guide%2C+University+of+California%2C+Los+Angeles.+&btnG=

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03935035/Prot_SAP_000.pdf
  • Informed Consent Form: Assent Form for participants aged 12-15 (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03935035/ICF_001.pdf
  • Informed Consent Form: Consent Form for participants aged 16-17 (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03935035/ICF_002.pdf
  • Informed Consent Form: Parental consent form for parental participation (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03935035/ICF_003.pdf
  • Informed Consent Form: Parental consent form for participants aged 12-15 (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03935035/ICF_004.pdf